CLINICAL TRIAL: NCT07227571
Title: FIERCe: FOLR1 Immune Effector Cell Therapy Against Advanced Osteosarcoma
Brief Title: Genetically Engineered Cells (FH-FOLR1 ST CAR T Cells) for the Treatment of Advanced Refractory or Recurrent/Progressive Osteosarcoma, FIERCe Trial
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Washington Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1125765; NCI-2025-08064 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FH20941 (Other: Fred Hutch/University of Washington/Seattle Children's Cancer Consortium)
Record Dates: First submitted 2025-11-10; First posted 2025-11-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Advanced Osteosarcoma; Recurrent Osteosarcoma; Refractory Osteosarcoma
Keywords: Bones and Joints
MeSH Terms: conditions — Osteosarcoma | interventions — Leukapheresis; fludarabine; Cyclophosphamide; Magnetic Resonance Spectroscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (FH-FOLR1 ST CAR T cells) (Experimental): Patients undergo leukapheresis for manufacturing of the FH-FOLR1 ST CAR T cell product on study. Patients will receive lymphodepleting therapy with fludarabine IV on days -5 to -2 and cyclophosphamide IV on days -3 to -2. Patients receive FH-FOLR1 ST CAR T cells IV on day 0, 1 or 2 in the absence of unacceptable toxicity. Patients also undergo echocardiography or multigated acquisition scan (MUGA), blood sample collection, and CT, MRI or PET throughout the study. Additionally, patients may have the option of undergoing tumor biopsy on study.
  Interventions: Biological: FH FOLR1 ST CAR T-cells; Procedure: Leukapheresis; Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Biopsy Procedure

INTERVENTIONS:
Biological: FH FOLR1 ST CAR T-cells — Given IV
  Other Names: Anti-FOLR1 CAR-T Cells; FH-FOLR1 CAR T Cells
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocyte Adsorptive Apheresis; Leukocytopheresis; Therapeutic Leukopheresis; White Blood Cell Reduction Apheresis
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Cyclophosphamide — Given IV
  Other Names: Cytoxan; Neosar; Revimmune; Cycloblastin
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide ventriculography
Procedure: Biospecimen Collection — Undergo blood sample collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CT; CT Scan; CAT Scan; Computed Axial Tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: PET; PET Scan
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Bx

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of FH-FOLR1 ST chimeric antigen receptor (CAR) T cells and how well they work in treating patients with osteosarcoma that recurred or spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) and that has not responded to previous treatment (refractory) or has come back after a period of improvement (recurrent)/is growing, spreading, or getting worse (progressive). CAR T-cell therapy is a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they attack tumor cells. T cells are taken from a patient's blood through a process called apheresis. Then the gene for a special receptor that binds to a certain protein on the patient's tumor cells, such as FOLR1, is added to the T cells in the laboratory. The special receptor is called a CAR. Large numbers of the CAR T cells are grown in the laboratory and given to the patient by an intravenous infusion. Chemotherapy drugs, such as fludarabine and cyclophosphamide, are given to a patient before the manufactured FH-FOLR1 ST CAR T cells to make room for the CAR T cells in the blood and to enhance the CAR T cell activity in the patient. FH-FOLR1 ST CAR T cells may be safe, tolerable, and/or effective in treating patients with advanced refractory or recurrent/progressive osteosarcoma.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of FH-FOLR1 ST CAR T cells.

Patients undergo leukapheresis for manufacturing of the FH-FOLR1 ST CAR T cell product on study. Patients receive lymphodepleting therapy with fludarabine intravenously (IV) on days -5 to -2 and cyclophosphamide IV on days -3 to -2. Patients receive FH-FOLR1 ST CAR T cells IV on day 0, 1 or 2 in the absence of unacceptable toxicity. Patients also undergo blood sample collection, and computed tomography (CT), magnetic resonance imaging (MRI) or positron emission tomography (PET) throughout the study. Additionally, patients have the option to undergo tumor biopsy on study. Patients will be monitored closely for at least 28 days after receiving CAR T cells.

After completion of study treatment, patients are followed up at days 1, 7, 14, 21, 28, and 42, months 2, 3, 6, 12, and 24, then every 6 months for 3 years followed by annually for 10 years. Patients with ongoing FH-FOLR1 ST CAR T cell persistence are also followed up in months 4, 5, 7, 8, 9, 10, 11, 15, and 18.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-75 years at the time of enrollment
* Tissue confirmation of osteosarcoma diagnosis
* Must have received an anthracycline-based regimen or been deemed ineligible to receive this therapy
* Must have at least one of the following in the 6 months prior to trial consent:

  * New site of measurable disease by radiographic imaging or histologic confirmation
  * New site of evaluable disease by radiographic imaging or histologic confirmation
  * Greater than 20% increase in at least one tumor dimension documented by CT/MRI, AND a minimum absolute increase of 5 mm in longest dimension of existing lesion(s) (previously irradiated lesions may be included)
  * Persistent measurable disease or fludeoxyglucose F-18 (FDG)-PET avid bone metastasis that has failed to achieve complete remission to upfront conventional therapy (surgery, radiotherapy, and/or chemotherapy)
* All anti-cancer therapy must be discontinued at enrollment/time of apheresis, with the following washout periods observed:

  * Chemotherapy and biologic agents: ≥ 7 days prior to enrollment
  * Steroid use: All corticosteroid therapy (unless physiologic replacement dosing and/or topical administration (e.g., inhaled or dermatologic) ≥ 7 days prior to enrollment
  * Tyrosine kinase inhibitor (TKI) use: ≥ 7 days prior to enrollment
  * Antitumor antibody therapy (including immune checkpoint inhibitor) must be ≥ 3 half-lives or 30 days, whichever is shorter, from time of enrollment
  * FOLR1 targeting therapy must be discontinued at least 30 days prior to enrollment
  * Gene modified cellular therapy: At enrollment, must be at least 30 days from most recent gene modified cell therapy infusion and document no evidence of modified cells in the peripheral blood OR must be at least 60 days from most recent gene modified cell therapy
  * Washout periods not applicable to patients with apheresis product or usable T cell product available for use at time of enrollment
* Potential trial participants should have recovered to grade 1 from clinically significant adverse events of their most recent therapy/intervention prior to enrollment
* Ability to understand and willingness to sign a written informed consent document.
* Females of child-bearing potential and fertile male participants must be willing to use an effective contraceptive method before, during, and for at least 12 months after the FOLR1 CART cell infusion
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (if treated at adult facility) or Lansky/Karnofsky score ≥ 60 (if treated at pediatric facility). Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for purposes of assessing performance status
* Life expectancy ≥ 8 weeks
* Able to tolerate apheresis, including placement of temporary apheresis catheter, if necessary, or already has an apheresis product available for use in manufacturing
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Participants with treated brain metastases are eligible if they meet the following criteria:

  * Follow-up brain imaging taken at screening demonstrates no evidence of progression and that imaging occurs 3 months after central nervous system (CNS)-directed therapy has been completed
  * No ongoing, symptomatic CNS pathology requiring medical intervention
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN) based on age and gender; or estimated creatinine clearance > 50 mL/min as calculated using the Cockcroft-Gault formula and not dialysis dependent

  * Age: 1 to < 2 years; maximum serum creatinine (mg/dL): 0.6 (male), 0.6 (female)
  * Age: 2 to < 6 years; maximum serum creatinine (mg/dL): 0.8 (male), 0.8 (female)
  * Age: 6 to < 10 years; maximum serum creatinine (mg/dL): 1 (male), 1 (female)
  * Age: 10 to < 13 years; maximum serum creatinine (mg/dL): 1.2 (male), 1.2 (female)
  * Age: 13 to < 16 years; maximum serum creatinine (mg/dL): 1.5 (male), 1.4 (female)
  * Age: ≥ 16 years; maximum serum creatinine (mg/dL): 1.7 (male), 1.4 (female)
* Total bilirubin ≤ 3 x ULN or conjugated bilirubin ≤ 2 mg/dL. Participants with suspected Gilbert syndrome may be included if total bilirubin (Bili) > 3 mg/dL but no other evidence of hepatic dysfunction
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 5 x ULN
* Pulmonary: ≤ grade 1 dyspnea at rest and arterial oxygen saturation (SaO2) ≥ 92% on ambient air. If pulmonary function tests (PFTs) are performed based on the clinical judgement of the treating physician, participants with forced expiratory volume in 1 second (FEVI) ≥ 50% of predicted and diffusion capacity of the lung for carbon monoxide (DLCO) (corrected) of ≥ 40% of predicted will be eligible
* Left ventricular ejection fraction (LVEF) may be established with echocardiogram or MUGA scan, and left ejection fraction must be ≥ 50% or shortening fraction ≥ 28%
* Absolute neutrophil count (ANC) ≥ 500 cells/ mm^3
* Hemoglobin ≥ 8 g/dL
* Platelets ≥ 100,000 per mm^3
* Participants receiving blood product transfusion are acceptable as long as they are not determined to be transfusion refractory

Exclusion Criteria:

* Active autoimmune disease: Participants with active autoimmune disease requiring immunosuppressive therapy are excluded. Case by case exemptions are possible with approval by PI
* Corticosteroid therapy at a dose equivalent of > 15 mg of prednisone per day (or equivalent). Pulsed corticosteroid use for disease control is acceptable. For participants weighing ≤ 30 kg, systemic steroids ≥ 0.5 mg prednisone equivalent/kg/day
* Concurrent use of other investigational anti-cancer agents
* Active uncontrolled infection: HIV positive participants on highly active antiretroviral therapy (HAART) with a CD4 count > 500 cells/mm^3 are considered controlled, as are individuals with a history of hepatitis C who have successfully completed antiviral therapy with an undetectable viral load, and those with hepatitis B who have hepatitis well controlled on medication
* Uncontrolled concurrent illness: Participants may not have uncontrolled or concurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia that would limit compliance with study requirements
* Active treatment for prior immune related adverse event to any immunotherapy: Participants receiving ongoing treatment for prior serious immune-related adverse events are excluded, with exception of hormone supplementation or corticosteroid therapy at equivalent of > 15 mg prednisone (or equivalent) per day, unless otherwise approved by PI
* Significant underlying neurologic disease: Study participants must not have significant active underlying neurologic disease, unless approved by PI. Peripheral neuropathy related to diabetes or prior chemotherapy is acceptable
* Pregnant, possibly pregnant or those expecting to conceive or father children for the duration of the trial through 4 months after T cell infusion
* Participants unwilling to provide consent/assent for participation in the study and 15-year follow-up period if CAR T cell therapy is administered
* Other medical, social, or psychiatric factor that interferes with medical appropriateness and/or ability to comply with study, as determined by the PI
* Known allergic reactions to any of the components of study treatments

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2044-01-31 (Estimated); Study Completion 2044-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related unexpected grade 3 or higher toxicity | Up to 28 days post infusion
Maximum tolerated dose/recommended phase 2 dose | Up to 28 days post infusion
  Will be defined as the highest T cell dose from among those tested for which the dose limiting toxicity (DLT) rate is closest to 28% and that at least 4 participants have been evaluated at that level. All observed DLT outcomes for toxicity-evaluable participants will be tabulated by dose level. Will employ a novel Bayesian optimal interval design.

SECONDARY OUTCOMES:
Progression free survival | From initiation of protocol treatment to disease progression or death of any cause, assessed up to 1 year post infusion
Overall survival | From initiation of protocol treatment to death of any cause, assessed up to 1 year post infusion
Overall response rate (ORR) | Up to 1 year post infusion
  Will be defined as complete response and partial response per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
Stable disease (SD) rate | Up to 1 year post infusion
  Will be evaluated using RECIST 1.1 criteria.
Clinical benefit rate | Up to 1 year post infusion
  Will be defined as ORR plus SD by RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Choe, MD, Principal Investigator — Fred Hutch/University of Washington/Seattle Children's Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington/Seattle Children's Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No